CLINICAL TRIAL: NCT03533725
Title: Breastfeeding Education Support Tool for Baby
Acronym: BEST4Baby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Jawaharlal Nehru Medical College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17F.517
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Breastfeeding
Keywords: Initiation, Exclusivity, Duration
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Intervention group having peer counseling and education and a comparative (control) group having standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Breastfeeding counseling and education services using mHealth tools
  Interventions: Other: Breastfeeding counseling and education services
- Comparative control group (No Intervention): No intervention, only standard of care

INTERVENTIONS:
Other: Breastfeeding counseling and education services — Breastfeeding counseling and education by educated and trained peer counselors using mHealth tools
  Arms: Intervention group

SUMMARY:
This study will compare data associated with breastfeeding experiences and outcomes--specifically, breastfeeding continuation after initiation, exclusivity for 6 months of an infant's life, and breastfeeding duration--among 120 subjects recruited late in pregnancy and provided peer counseling and education services incorporating mobile health (mHealth) tools during a period of at least 6 months post-delivery with the data collected from a control group of approximately 120 mothers that did not receive the study intervention.

DETAILED DESCRIPTION:
Approximately 24 women that are experienced in breastfeeding will be recruited to serve in the role of breastfeeding peer counselors. These women will assess usability and acceptability of mobile health (mHealth) education tools designed following a series of focus groups for the project, Breastfeeding Education Support Tool for Baby. The mHealth tools will be used during the training and education of the peer counselor subjects. Following appropriate modification, some of the mHealth tools will be used with a total of approximately 120 women recruited late in pregnancy for initial breastfeeding counseling before delivery and the subsequent provision, for at least 6 months post-delivery, of home visits for peer counseling and education that integrates use of mHealth tools. Peer counselors and research staff will gather data from mothers receiving the intervention about breastfeeding experiences and outcomes, including breastfeeding continuation after initiation, exclusivity for 6 months of an infant's life, and breastfeeding duration. This data will be compared to data obtained through surveys administered to a control group of approximately 120 maternal subjects that received standard pre- and post-delivery care but not the study intervention of peer counseling and education using mHealth tools.

ELIGIBILITY:
A. Peer counselors

Inclusion Criteria:

Personal experience with breastfeeding - Residence in an intervention cluster

Exclusion Criteria:

- Failing to participate in peer counselor education/training provided for the study

B. Intervention Pregnant women-mothers

Inclusion Criteria:

* Willingness to consent to assignment to a breastfeeding peer counselor and to participate in counseling and education visits
* Residence in an intervention cluster and intent to remain in the intervention area for a minimum of 6 months post-delivery

Exclusion Criteria:

- Pregnant women-mothers that indicate before delivery that they will not initiate breastfeeding

C. Control Subjects

Inclusion Criteria:

* Mothers delivering during the study period that live in a non-intervention area that has been designated for recruitment of control subjects
* Willingness to participate in a survey enabling collection of data for comparative purposes

Exclusion Criteria:

- None

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females as study involves an activity only females can perform and only females could be considered peers of mothers
Enrollment: 247 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding initiation soon after birth | Ideally within an hour following a normal delivery
  Maternal subjects' compliance with the recommendation to initiate breastfeeding soon after delivery
Exclusivity of breastfeeding during the first 6 months following an infant's birth | First 6 months following an infant's birth
  Maternal subjects' compliance with the recommendation to provide only breast milk
Breastfeeding continuation (along with supplemental feeding) after an infant reaches 6 months of age | As the study is time-limited, assessment will occur 6-9 months following an infant's birth
  Maternal subjects' compliance with the recommendation for continued breastfeeding along with supplemental feeding after an infant reaches 6 months of age

SECONDARY OUTCOMES:
Usability rating of the mHealth tools by peer counselors post-training | At the end of counseling education/training (project months 8-9)
  Peer counselors will complete a scale, mHealth Tools Usability Scale for Peer Counselors
  Information relevant to this scale:
  Likert scale with 10 statements associated with usability: 5 positive and 5 negative
  Range of responses 1. Strongly Disagree, 2. Disagree, 3. Neutral/No Opinion, 4. Agree, 5. Strongly Agree
  Scoring: For positive items, the score contribution is the scale position number minus 1; and for negative items the contribution is 5 minus the scale position number. All scores are totaled and multiplied by 2.5, resulting in a total score per subject of 0-100. With this scoring method the higher the score, the greater is usability of the mHealth tools as perceived by the peer counselors after training but before actual use with mothers.
  Scale is based upon one initially developed and tested by Digital Equipment Corporation; items have been slightly modified to achieve a better match with the BEST4Baby pilot.
Usability rating of the mHealth tools by peer counselors based on use with mothers | Once peer counselors complete delivery of services to assigned maternal subjects (by months 22-23 of the project)
  Peer counselors will complete a scale, mHealth Tools Usability Scale for Peer Counselors Based Upon Use with Mothers
  Information relevant to the scale:
  Likert Scale with 10 statements associated with usability: 5 positive and 5 negative
  Range of responses 1. Strongly Disagree, 2. Disagree, 3. Neutral/No Opinion, 4. Agree, 5. Strongly Agree
  Scoring: For positive items, the score contribution is the scale position number minus 1; and for negative items the contribution is 5 minus the scale position number. All scores are totaled and multiplied by 2.5, resulting in a total score per subject of 0-100. With this scoring method the higher the score, the greater is usability of the mHealth tools.as perceived by peer counselors based upon use with the mothers.
  The scale is similar to the one for Secondary Outcome Measure 4 (and is similar to the referenced Digital Equipment Corporation scale).
Acceptability rating of BEST4Baby program features by mothers | 3 months post-delivery
  Maternal subjects will utilize a scale, Mothers Acceptability Rating Scale for BEST4Baby Program Features
  Information relevant to this scale:
  Likert Scale with 10 statements associated with features of the BEST4Baby program: 5 positive and 5 negative (related to peer counselor, home visits, educational modality, etc.)
  Range of responses 1. Very unacceptable, 2. Unacceptable, 3. Neutral/No Opinion, 4. Acceptable, 5. Very Acceptable
  Scoring: For positive items, the score contribution is the scale position number minus 1; and for negative items the contribution is 5 minus the scale position number. All scores are totaled and multiplied by 2.5, resulting in a total score per subject of 0-100. With this scoring method the higher the score, the more acceptable were program features to the maternal subject.
Satisfaction rating of mothers with BEST4Baby counseling and education services as delivered | 6-9 months post-delivery
  Maternal subjects will complete a scale, Mothers Level of Satisfaction with BEST4Baby Services as Delivered
  Information relevant to this scale:
  Likert Scale with 10 statements associated with level of satisfaction with BEST4Baby counseling and education services as delivered: 5 positive and 5 negative
  Range of responses 1. Very unsatisfied, 2. Unsatisfied, 3. Neutral/No Opinion, 4. Satisfied, 5. Very Satisfied
  Scoring: For positive items, the score contribution is the scale position number minus 1; and for negative items the contribution is 5 minus the scale position number. All scores are totaled and multiplied by 2.5, resulting in a total score per subject of 0-100. With this scoring method the higher the score, the more satisfied the subject was with the counseling and education services as delivered.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Derman, MD,, Principal Investigator — Thomas Jefferson University; Shivaprasad S. Goudar, MD, MHPE, Study Director — Jawaharlal Nehru Medical College, KLE Academy of Higher Education
Locations (1):
- Jawaharlal Nehru Medical College, Belagavi, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for the primary and secondary outcomes are expected to be shared in publications resulting from this pilot study.
Supporting Information: Study Protocol
Time Frame: Estimated availability : within 18 months of study closure.
Access Criteria: Global health researchers upon request

REFERENCES:
- [Result] Charantimath U, Bellad R, Majantashetti N, Washio Y, Derman R, Kelly PJ, Short V, Chung E, Goudar S. Facilitators and challenges to exclusive breastfeeding in Belagavi District, Karnataka, India. PLoS One. 2020 May 4;15(5):e0231755. doi: 10.1371/journal.pone.0231755. eCollection 2020. PMID 32365108
- [Result] Short VL, Bellad RM, Kelly PJ, Washio Y, Ma T, Chang K, Majantashetti NS, Charantimath US, Jaeger FJ, Lalakia P, Goudar SS, Derman R. Feasibility, acceptability, and preliminary impact of an mHealth supported breastfeeding peer counselor intervention in rural India. Int J Gynaecol Obstet. 2022 Jan;156(1):48-54. doi: 10.1002/ijgo.13599. Epub 2021 Feb 20. PMID 33454986
- [Derived] Ma T, Chang K, Alyusuf A, Bajracharya E, Washio Y, Kelly PJ, Bellad RM, Mahantashetti NS, Charantimath U, Short VL, Lalakia P, Jaeger F, Goudar S, Derman R. Design, Development, and Testing of BEST4Baby, an mHealth Technology to Support Exclusive Breastfeeding in India: Pilot Study. JMIR Form Res. 2022 Sep 8;6(9):e32795. doi: 10.2196/32795. PMID 36074546

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT03533725/Prot_SAP_000.pdf
  • Informed Consent Form: BEST4 Baby Consent--Peer Counselors (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03533725/ICF_001.pdf
  • Informed Consent Form: BEST4Baby Consent--Participants (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03533725/ICF_002.pdf